CLINICAL TRIAL: NCT05235659
Title: Empowering Youth in Care Against (re-)Victimization (Subproject 4): A Randomized Balanced Factorial Trial Examining an Internet-based Prevention Program for Primary Caregivers
Brief Title: EMPOWERYOU: Examining an Internet-based Prevention Program for Primary Caregivers
Acronym: EMPOWERYOU-4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bremen (Other)
Collaborators: RWTH Aachen University (Other); Bielefeld University (Other); Medical School Berlin (Other); Karlsruhe Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: UBremen; FKZ 01KR1806D (Other Grant/Funding Number: German Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2022-01-27; First posted 2022-02-11 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Victimisation
Keywords: multiphase optimization strategy; foster children; parenting; revictimization; online-intervention

STUDY DESIGN:
Intervention Model Description: 2 x 2 x 2 x 2 full factorial design
Masking Description: Study staff at University of Bremen will not view the allocation sequence. The database will not reveal participants' treatment condition to study staff until after the family´s eligibility was verified (after pre-assessment). Families will be informed of their allocation status after baseline data collection is completed to assure that participants are blind to allocation during the initial assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules
- Condition 2 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental condition "My coach"
- Condition 3 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules and experimental module "Who am I and where do I belong?"
- Condition 4 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental modules "Who am I and where do I belong?" and "My coach"
- Condition 5 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules and experimental module "You are safe here"
- Condition 6 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental modules "You are safe here" and "My coach"
- Condition 7 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules and experimental modules "You are safe here" and "Who am I and where do I belong?"
- Condition 8 (Experimental): Component 1 (Watch out!): off, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental modules "You are safe here", "Who am I and where do I belong?", and "My coach"
- Condition 9 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules and experimental module "Watch out!"
- Condition 10 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental modules "Watch out!" and "My coach"
- Condition 11 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules and experimental modules "Watch out!" and "Who am I and where do I belong?"
- Condition 12 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): off, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental modules "Watch out!", "Who am I and where do I belong?", and "My coach"
- Condition 13 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules and experimental modules "Watch out!" and "You are safe here"
- Condition 14 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): off, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental modules "Watch out!", "You are safe here", and "My coach"
- Condition 15 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): off
  Interventions: Behavioral: Basic modules and experimental modules "Watch out!", "You are safe here", and "Who am I and where do I belong?"
- Condition 16 (Experimental): Component 1 (Watch out!): on, Component 2 ("You are safe here"): on, Component 3 ("Who am I and where do I belong?"): on, Component 4 ("My coach"): on
  Interventions: Behavioral: Basic modules and experimental modules "Watch out!", "You are safe here", "Who am I and where do I belong?", and "My coach"

INTERVENTIONS:
Behavioral: Basic modules — Caregivers will only have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child.
  Arms: Condition 1
Behavioral: Basic modules and experimental condition "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Professional support of the caregiver will be provided. Caregivers will receive one phone call (50 minutes) to support processing of information from module 1 and 2. Finally, they will receive text messages or emails with the core message of the modules.
  Arms: Condition 2
Behavioral: Basic modules and experimental module "Who am I and where do I belong?" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to the module 5 "Who am I and where do I belong?" This module will support caregivers in helping their child developing an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers.
  Arms: Condition 3
Behavioral: Basic modules and experimental modules "Who am I and where do I belong?" and "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to the module 5 "Who am I and where do I belong?" This module will support caregivers in helping their child developing an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers. Professional support of the caregiver will be provided. Caregivers will receive two phone calls (each 50 minutes) to support processing of information from module 1, 2, and 5. Finally, they will receive text messages or emails with the core message of the modules.
  Arms: Condition 4
Behavioral: Basic modules and experimental module "You are safe here" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 4 "You are safe here" to improve children´s relationship-related safety and facilitate solid relationships with family and peers.
  Arms: Condition 5
Behavioral: Basic modules and experimental modules "You are safe here" and "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 4 "You are safe here" to improve children´s relationship-related safety and facilitate solid relationships with family and peers. Professional support of the caregiver will be provided. Caregivers will receive two phone calls (each 50 minutes) to support processing of information from module 1, 2, and 4. Finally, they will receive text messages or emails with the core message of the modules.
  Arms: Condition 6
Behavioral: Basic modules and experimental modules "You are safe here" and "Who am I and where do I belong?" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 4 "You are safe here" to improve children´s relationship-related safety and facilitate solid relationships with family and peers. Caregivers will have access to the module 5 "Who am I and where do I belong?" This module will support caregivers in helping their child developing an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers.
  Arms: Condition 7
Behavioral: Basic modules and experimental modules "You are safe here", "Who am I and where do I belong?", and "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 4 "You are safe here" to improve children´s relationship-related safety and facilitate solid relationships with family and peers. Caregivers will have access to the module 5 "Who am I and where do I belong?" This module will support caregivers in helping their child developing an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers. Professional support of the caregiver will be provided. Caregivers will receive three phone calls (each 50 minutes) to support processing of information from module 1, 2, 4, and 5. Finally, they will receive text messages or emails with the core message of the modules.
  Arms: Condition 8
Behavioral: Basic modules and experimental module "Watch out!" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior.
  Arms: Condition 9
Behavioral: Basic modules and experimental modules "Watch out!" and "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior. Professional support of the caregiver will be provided. Caregivers will receive two phone calls (each 50 minutes) to support processing of information from module 1, 2, and 3. Finally, they will receive text messages or emails with the core message of the modules.
  Arms: Condition 10
Behavioral: Basic modules and experimental modules "Watch out!" and "Who am I and where do I belong?" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior. Caregivers will have access to the module 5 "Who am I and where do I belong?" This module will support caregivers in helping their child developing an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers.
  Arms: Condition 11
Behavioral: Basic modules and experimental modules "Watch out!", "Who am I and where do I belong?", and "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior. Caregivers will have access to the module 5 "Who am I and where do I belong?" This module will support caregivers in helping their child developing an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers. Professional support of the caregiver will be provided. Caregivers will receive three phone calls (each 50 minutes) to support processing of information from module 1, 2, 3, and 5. Finally, they will receive text messages or emails with the core message of the modules.
  Arms: Condition 12
Behavioral: Basic modules and experimental modules "Watch out!" and "You are safe here" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior. Caregivers will have access to module 4 "You are safe here" to improve children´s relationship-related safety and facilitate solid relationships with family and peers.
  Arms: Condition 13
Behavioral: Basic modules and experimental modules "Watch out!", "You are safe here", and "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior. Caregivers will have access to module 4 "You are safe here" to improve children´s relationship-related safety and facilitate solid relationships with family and peers. Professional support of the caregiver will be provided. Caregivers will receive three phone calls (each 50 minutes) to support processing of information from module 1, 2, 3, and 4. Finally, they will receive text messages or emails with the core message of the modules.
  Arms: Condition 14
Behavioral: Basic modules and experimental modules "Watch out!", "You are safe here", and "Who am I and where do I belong?" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation of caregiver and child. Caregivers will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior. Caregivers will have access to module 4 "You are safe here" to improve children´s relationship-related safety and facilitate solid relationships with family and peers. Caregivers will have access to the module 5 "Who am I and where do I belong?" This module will support caregivers in helping their child developing an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers.
  Arms: Condition 15
Behavioral: Basic modules and experimental modules "Watch out!", "You are safe here", "Who am I and where do I belong?", and "My coach" — Caregivers will have access to the two basic modules (1&2) in order to increase knowledge on parental self-care and facilitating the self-worth of the child as well as emotional regulation. They will have access to module 3 "Watch out!" on improving children´s relationship-related risk detection and self-protective behavior. Further access will be provided to module 4 "You are safe here" on improving children´s relationship-related safety and facilitating solid relationships. Access to module 5 "Who am I and where do I belong?" will support caregivers in helping their child develop an identity of their choice, while providing the freedom to consider potential contributing influences of the family of origin, foster family, and peers. Professional support will be provided. They will receive four phone calls (each 50 minutes) to support processing of information from module 1, 2, 3, 4, and 5. Text messages or emails with the core message of the modules will be provided.
  Arms: Condition 16

SUMMARY:
The primary aim of this study is to examine the effects of an internet-based prevention program for primary caregivers of preadolescent Youth in Care (Y-IC) on (re-)victimization. We aim to identify the most effective intervention components by using a randomized factorial design, based on the Multiphase Optimization Strategy (MOST; Collins, 2018). In a 2 x 2 x 2 x 2 factorial trial, an initial N = 317 foster caregivers with children ages 8 - 13 are randomly assigned to one of 16 conditions. The primary outcome is the rate of (re-)victimization from pre- to 3-month follow-up. Secondary outcomes include risk-taking and functional behaviors in relationships. All caregivers will receive access to all components after trial ends if there is no significant harm associated with any of the intervention component. Participants in the condition with all component levels on are expected to show the best improvement. Anticipated date for study completion is determined by the funding period. However, we plan to apply for a study extension.

DETAILED DESCRIPTION:
Given that childhood victimization leads to an increased vulnerability for subsequent revictimization in adolescence, findings highlight a strong need for evidence-based prevention programs targeting children with a history of child maltreatment as a high-risk population of revictimization. However, evidence-based programs for foster parents that aim to prevent revictimization of the child, while addressing the needs of the caregivers are scarce. In order to develop and tailor such services to foster parents (and youth in care) with maltreatment experiences, we developed a consumer-informed conceptual model in a prior project (EMPOWERYOU SP3) that outlines the key mediators which may impact upon the risk of revictimization and how we plan to address these with different intervention components. Thus, in subproject 3 the conceptual model and the online-intervention components were developed, involving the participants themselves as well as relevant stakeholders. The usability of the online-intervention and the feasibility of the clinical trial (EMPOWERYOU SP4) was piloted in subproject 3 (March 2021 - September 2021).

In subproject 4, we will conduct a factorial study to tear apart the main effects of each intervention component on the mediator and outcome of interest, including potential interaction effects. This will help optimizing the intervention approach. The full online-intervention comprises five content modules and a coach, who is supporting the caregiver with up to four phone-calls (50 minutes each) and short message service (SMS) or e-mail reminders. Caregivers have two weeks to work through one module. Every caregiver will receive the first two basic modules on parental self-care and child´s self-worth and emotional regulation. This allows us to offer some level of support in all conditions including the condition with the lowest component level across all factors.

Based on the MOST principles, this study will use a 2 x 2 x 2 x 2 full factorial design by randomly allocating families with equal probability to one of 16 experimental conditions. However, this factorial experiment does not represent a 16-arm randomized controlled trial (RCT). The ultimate goal is to choose from a set of four intervention components with two levels each (on/off) the one(s) that best reduce and prevent (re-)victimization. The following intervention components have been selected (three content components, one engagement/adherence component):

1. Component: "Watch out!" (on/off): Improving relationship-related risk detection and self-protective behavior
2. Component: "You are safe here" (on/off): Improving relationship-related safety and facilitating solid relationships
3. Component: "Who am I and where do I belong?" (on/off): Supporting the child constructing an identity
4. Component: "My Coach" (on/off): Professional support of the caregiver in form of up to four phone calls with a coach (i.e., one call per module 1&2 (combined), 3, 4, and 5).

The primary research objectives are:

1. To examine the efficacy of selected candidate components on primary outcome, the risk of re-victimization, at follow-up (i.e., 3 months post intervention; approx. 24 weeks after baseline)
2. To examine the efficacy of selected candidate components on secondary outcomes (risk-taking behavior and functional behavior in relationships with caregiver, siblings, peers, and others) at post-test (i.e., 1 week post intervention; approx. 12 weeks after baseline)

The secondary objectives are:

1. To test enduring effects of selected components on secondary outcomes at 3-month follow-up
2. To test mediating effects of theory-driven factors on the relationship between selected components on secondary outcomes
3. To explore whether there are any interaction effects between components on primary or secondary outcomes
4. To conduct exploratory analyses of potential moderators

Based on the conceptual model described above, this study will examine the following hypotheses related to the main effects of intervention components:

1. Component "Watch out!" - Relationship-related risks: We hypothesize that receiving this component will result in better detection of risk signals in relationships and less risk-taking cognitions. This will lead to less relationship-related risk-taking behavior which in turn will result in reductions of re-victimization experiences and others secondary outcomes.
2. Component "You are safe here" - Relationship-related safety: We hypothesize that receiving this component will result in better detection of safety signals in relationships and more emotional security. This will lead to more functional relationship behavior which in turn will result in reductions of (re-)victimization experiences and other secondary outcomes.
3. Component "Who am I and where do I belong?" - Constructing identity: We hypothesize that receiving this component will increase parental support in the child´s constructing of identity. This will lead to a more positive self-appraisal and in turn to less risk-taking and more functional relationship behavior, which in turn will result in reductions of (re-)victimization experiences and other secondary outcomes.
4. Component "My Coach" - Professional support: We hypothesize that professional support from a parent coach who is facilitating each component, will result in higher program adherence/engagement which will yield larger intervention effects on primary and secondary outcomes than without professional support.
5. We hypothesize that there will be an interaction effect between the relationship risk and relationship safety components. When both components will be present, the effect will be larger compared to only one of them present.
6. We hypothesize that there will be an interaction effect between each component and the professional support component, such that with professional support, the effects of each component will be larger than without professional support via greater adherence/engagement of the caregiver.

ELIGIBILITY:
Inclusion Criteria:

- primary caregivers (foster or adoptive) of children aged 8 to 13 years old

Exclusion Criteria:

* acute child endangerment
* short-term foster families ("Bereitschaftspflege")
* family care ("Verwandschaftspflege")
* insufficient German language knowledge

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 317 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of (re-)victimization | Pre and 3 months post intervention; approx. 24 weeks after baseline
  The (re-)victimization composite score derived from two parent-report measures: The Juvenile Victimization Questionnaire (JVQ) and the Bullying screener. The JVQ is a widely used measure to assess victimization in children aged 8 to 17 years. It consists of 37 items spanning five domains: crime, child maltreatment, peer and sibling victimization, sexual victimization and witnessing crime with follow-up questions that also assess the frequency and perpetrators of the victimization events. Caregivers will be asked whether the child was exposed to the respective event during life and (if yes) during the last 3 months. Participants respond with yes (1) or no (0). The Bullying screener is a 6-item screening tool. After the respective definition of bullying type, caregivers are asked how often these things happened to the child or how often he/she has done this to others in the last 3 months. Caregivers then respond on a 4-point scale from never to a lot (at least once a week).

SECONDARY OUTCOMES:
Change in frequency of relationship-related risk-taking behavior | Pre and 1 week post intervention; approx. 12 weeks after baseline
  Relationship-related risk-taking behaviors wilt be assessed with a self-developed questionnaire on risk situations in relationships. The questionnaire comprises 14 risky situations (e.g., "How often has someone done something to your child even though he/she did not want that and said "no"?"). Caregivers and children are asked how often the risky situation occurred during the last three months (frequency).
Change in level of functional behavior in relationship with caregiver | Pre and 1 week post intervention; approx. 12 weeks after baseline
  To assess functional relationship behavior in the relationship with the caregiver, the subscales communication and involvement of the Parenting Relationship Questionnaire (PRQ) will be used (22 items).
Change in level of functional behavior in relationship with siblings | Pre and 1 week post intervention; approx. 12 weeks after baseline
  To assess functional relationship behavior in relationship with siblings, we will use the seven subscales referring to "warmth and closeness" of the Sibling Relationship Questionnaires (SRQ-deu; 21 items).
Change in level of functional behavior across unspecified relationships | Pre and 1 week post intervention; approx. 12 weeks after baseline
  To assess functional relationship behavior across unspecified relationships, the Relationship Problems Questionnaire (RPQ) will be used (10 items).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Heinrichs, Prof. Dr., Principal Investigator — University of Bremen; Kerstin Konrad, Prof. Dr., Principal Investigator — RWTH Aachen University; Arnold Lohaus, Prof. Dr., Principal Investigator — Bielefeld University; Birgit Wagner, Prof. Dr., Principal Investigator — Medical School Berlin; Ulrich Eber-Priemer, Prof. Dr., Principal Investigator — Karlsruhe Institute of Technology
Locations (2):
- Germany (2):
  - Bielefeld University, Bielefeld
  - University of Bremen, Bremen

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share results with members of the scientific community. The anonymized data set will be stored for 10 years and shared with other research teams upon request, using a repository that will be chosen by the consortium (advised by the DSMB).
Supporting Information: Study Protocol
Time Frame: IPD will be shared after data analysis and dissemination of main findings. Study Protocol will be shared once it is published (preferably open access). The clinical trial registry is mirroring the study protocol and includes excerpts of the submitted manuscript.
Access Criteria: The anonymized data set will be shared with other research teams upon request.

REFERENCES:
- [Derived] Heinrichs N, Bruhl A. Preventing Revictimization Through a Web-Based Intervention for Primary Caregivers of Youth in Care (EMPOWERYOU): Protocol for a Randomized Factorial Trial. JMIR Res Protoc. 2022 Oct 24;11(10):e38183. doi: 10.2196/38183. PMID 36279162
- See also: Study website (for subproject 4) — http://empoweryou-programm.de